CLINICAL TRIAL: NCT05582135
Title: Epidural Esketamine and Morphine for Postoperative Analgesia After Caesarean Delivery: A Pilot Study
Brief Title: Postoperative Analgesic Effect of Esketamine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanhan County People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XuanhanCo
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Gynecological; Surgery (Previous), Affecting Fetus or Newborn, Due to Obstructed Labor; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Morphine; Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group A (Active Comparator): The parturients in group A were administered 2 mg morphine sulfate through the epidural catheter.
  Interventions: Drug: 2 mg morphine sulfate
- group B (Active Comparator): The parturients in group B were administered 0.25mg/kg of esketamine.
  Interventions: Drug: 0.25mg/kg esketamine
- group C (Active Comparator): The parturients in group C were administered 0.25mg/kg of esketamine in combination with 2 mg morphine sulfate.
  Interventions: Drug: 0.25mg/kg of esketamine in combination with 2 mg morphine sulfate
- group D (Active Comparator): The parturients in group D were administered 0.25mg/kg of esketamine in combination with 1 mg morphine sulfate.
  Interventions: Drug: 0.25mg/kg of esketamine in combination with 1 mg morphine sulfate

INTERVENTIONS:
Drug: 2 mg morphine sulfate — The parturients were administered 2 mg morphine sulfate through the epidural catheter. Sterile saline was added to make a total volume of 8 mL.
  Arms: group A
Drug: 0.25mg/kg esketamine — The parturients were administered 0.25mg/kg of esketamine through the epidural catheter. Sterile saline was added to make a total volume of 8 mL.
  Arms: group B
Drug: 0.25mg/kg of esketamine in combination with 2 mg morphine sulfate — The parturients were administered 0.25mg/kg of esketamine in combination with 2 mg morphine sulfate through the epidural catheter. Sterile saline was added to all combinations of the analgesic drugs to make a total volume of 8 mL.
  Arms: group C
Drug: 0.25mg/kg of esketamine in combination with 1 mg morphine sulfate — The parturients were administered 0.25mg/kg of esketamine in combination with 1 mg morphine sulfate through the epidural catheter. Sterile saline was added to all combinations of the analgesic drugs to make a total volume of 8 mL.
  Arms: group D

SUMMARY:
The aim of this study was to determine whether the addition of esketamine to morphine would improve postoperative analgesia after caesarean section.

Parturients who planned for a caesarean delivery using combined spinal-epidural anaesthesia with a request for postoperative anaesthesia were randomly divided into four groups (A, B, C and D). When the surgery was completed, the parturients in groups A, B, C and D were administered 2 mg morphine, 0.25mg/kg of esketamine, 0.25mg/kg of esketamine plus 2 mg morphine sulfate and 0.25mg/kg of esketamine plus 1 mg morphine through the epidural catheters, respectively. The postoperative pain at rest, pain with movement, the number of rescue analgesics and adverse effects were evaluated for 48 h after caesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous parturients who scheduled for elective caesarean delivery under spinal-epidural anaesthesia;
* parturients who had requested postoperative analgesia;
* parturients aged between 20-35 years old;
* parturients who had a full-term pregnancy;
* parturients who were identified as having a singleton pregnancy; and
* parturients who were categorised as having an American Society of Anaesthesiologists (ASA) physical status

Exclusion Criteria:

* parturients with severe internal, surgical or obstetric comorbidities (including spinal deformities, hypertension, placental abruption, cholestasis in pregnancy, asthma, heart disease and abnormal coagulation parameters)
* parturients with a known allergy to the drugs used in this study
* parturients with severe mental illness who could not comply with doctors' instructions
* parturients with chronic pain syndrome, which is defined as pain that persists for a period longer than 3 months

Ages: 20 Years to 32 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score at rest | Two hours after caesarean delivery
  The pain scores at rest were evaluated by the parturients themselves using a VAS based on a linear scale from 0 to 10, where 0 represented an absence of pain and 10 represented maximal pain.
Postoperative pain score at rest | Four hours after caesarean delivery
  The pain scores at rest were evaluated by the parturients themselves using a VAS based on a linear scale from 0 to 10, where 0 represented an absence of pain and 10 represented maximal pain.
Postoperative pain score at rest | Eight hours after caesarean delivery
  The pain scores at rest were evaluated by the parturients themselves using a VAS based on a linear scale from 0 to 10, where 0 represented an absence of pain and 10 represented maximal pain.
Postoperative pain score at rest | Twelve hours after caesarean delivery
  The pain scores at rest were evaluated by the parturients themselves using a VAS based on a linear scale from 0 to 10, where 0 represented an absence of pain and 10 represented maximal pain.
Postoperative pain score at rest | Twenty-four hours after caesarean delivery
  The pain scores at rest were evaluated by the parturients themselves using a VAS based on a linear scale from 0 to 10, where 0 represented an absence of pain and 10 represented maximal pain.
Postoperative pain score at rest | Forty-eight hours after caesarean delivery
  The pain scores at rest were evaluated by the parturients themselves using a VAS based on a linear scale from 0 to 10, where 0 represented an absence of pain and 10 represented maximal pain.
Postoperative pain score with movement | Two hours after caesarean delivery
  The pain scores on movement were evaluated by the parturients themselves using a VAS based on a linear scale from 0 to 10, where 0 represented an absence of pain and 10 represented maximal pain.
Postoperative pain score with movement | Four hours after caesarean delivery
  The pain scores on movement were evaluated by the parturients themselves using a VAS based on a linear scale from 0 to 10, where 0 represented an absence of pain and 10 represented maximal pain.
Postoperative pain score with movement | Eight hours after caesarean delivery
  The pain scores on movement were evaluated by the parturients themselves using a VAS based on a linear scale from 0 to 10, where 0 represented an absence of pain and 10 represented maximal pain.
Postoperative pain score with movement | Twelve hours after caesarean delivery
  The pain scores on movement were evaluated by the parturients themselves using a VAS based on a linear scale from 0 to 10, where 0 represented an absence of pain and 10 represented maximal pain.
Postoperative pain score with movement | Twenty-four hours after caesarean delivery
  The pain scores on movement were evaluated by the parturients themselves using a VAS based on a linear scale from 0 to 10, where 0 represented an absence of pain and 10 represented maximal pain.
Postoperative pain score with movement | Forty-eight hours after caesarean delivery
  The pain scores on movement were evaluated by the parturients themselves using a VAS based on a linear scale from 0 to 10, where 0 represented an absence of pain and 10 represented maximal pain.
number of rescue analgesics required | within Forty-eight hours of surgery
  The number of rescue analgesics required within 48 h of surgery was recorded

SECONDARY OUTCOMES:
systolic blood pressure (SBP) | Two hours after caesarean delivery
  Patient's systolic blood pressure (SBP)
systolic blood pressure (SBP) | Four hours after caesarean delivery
  Patient's systolic blood pressure (SBP)
systolic blood pressure (SBP) | Eight hours after caesarean delivery
  Patient's systolic blood pressure (SBP)
systolic blood pressure (SBP) | Twelve hours after caesarean delivery
  Patient's systolic blood pressure (SBP)
systolic blood pressure (SBP) | Twenty-four hours after caesarean delivery
  Patient's systolic blood pressure (SBP)
systolic blood pressure (SBP) | Forty-eight hours after caesarean delivery
  Patient's systolic blood pressure (SBP)
diastolic blood pressure (DBP) | Two hours after caesarean delivery
  Patient's diastolic blood pressure (DBP)
diastolic blood pressure (DBP) | Four hours after caesarean delivery
  Patient's diastolic blood pressure (DBP)
diastolic blood pressure (DBP) | Eight hours after caesarean delivery
  Patient's diastolic blood pressure (DBP)
diastolic blood pressure (DBP) | Twelve hours after caesarean delivery
  Patient's diastolic blood pressure (DBP)
diastolic blood pressure (DBP) | Twenty-four hours after caesarean delivery
  Patient's diastolic blood pressure (DBP)
diastolic blood pressure (DBP) | Forty-eight hours after caesarean delivery
  Patient's diastolic blood pressure (DBP)
heart rate (HR) | Two hours after caesarean delivery
  Patient's heart rate (HR)
heart rate (HR) | Four hours after caesarean delivery
  Patient's heart rate (HR)
heart rate (HR) | Eight hours after caesarean delivery
  Patient's heart rate (HR)
heart rate (HR) | Twelve hours after caesarean delivery
  Patient's heart rate (HR)
heart rate (HR) | Twenty-four hours after caesarean delivery
  Patient's heart rate (HR)
heart rate (HR) | Forty-eight hours after caesarean delivery
  Patient's heart rate (HR)
Blood oxygen saturation (SpO2) | Two hours after caesarean delivery
  Measurement of pulse Blood oxygen saturation (SpO2) in parturients
Blood oxygen saturation (SpO2) | Four hours after caesarean delivery
  Measurement of pulse Blood oxygen saturation (SpO2) in parturients
Blood oxygen saturation (SpO2) | Eight hours after caesarean delivery
  Measurement of pulse Blood oxygen saturation (SpO2) in parturients
Blood oxygen saturation (SpO2) | Twelve hours after caesarean delivery
  Measurement of pulse Blood oxygen saturation (SpO2) in parturients
Blood oxygen saturation (SpO2) | Twenty-four hours after caesarean delivery
  Measurement of pulse Blood oxygen saturation (SpO2) in parturients
Blood oxygen saturation (SpO2) | Forty-eight hours after caesarean delivery
  Measurement of pulse Blood oxygen saturation (SpO2) in parturients
Adverse events | within Forty-eight hours of surgery
  Adverse events that occurred after the administration of study drugs were also recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Qijun Ran, Dazhou, Sichuan, China